CLINICAL TRIAL: NCT05901662
Title: Older Volunteers' Competence Training for Community-based Long-term Care Services
Brief Title: Older Volunteers' Competence Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University (Other)
Responsible Party: Principal Investigator, Kuei-Min Chen, Ph.D., RN., Professor, Kaohsiung Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: KMUHIRB-E(I)-20220056
Record Dates: First submitted 2023-06-05; First posted 2023-06-13 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Volunteers
Keywords: knowledge and skills; motivation; self-efficacy; satisfaction
MeSH Terms: conditions — Personal Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Competence training program (Experimental): This group received a 3-hour weekly course training session in four consecutive weeks and provided services to community-dwelling older adults for two months.
  Interventions: Other: Competence training program
- Control (Active Comparator): This group provided their routine services at senior activity centers.
  Interventions: Other: Control

INTERVENTIONS:
Other: Competence training program — A 3-hour weekly course training session in four consecutive weeks and provided services to community-dwelling older adults for two months.
  Arms: Competence training program
Other: Control — This group provided their routine services at senior activity centers.
  Arms: Control

SUMMARY:
This project was aimed to evaluate the effectiveness of the competence training program in improving the knowledge and skills of volunteer work, the motivation for volunteering, self-efficacy, and satisfaction with volunteer work among older volunteers.

DETAILED DESCRIPTION:
A cluster-randomized controlled trial was conducted to test the effects of a 3-month comprehensive competence training program in improving the knowledge and skills of volunteer work, the motivation for volunteering, self-efficacy, and satisfaction with volunteer work among older volunteers. Using convenience sampling, 10 senior activity centers with 162 older volunteers were recruited and cluster-randomized to the intervention group (5 centers) or wait-list comparison group (5 centers). The intervention group received a 3-hour weekly course training session in four consecutive weeks and provided services to community-dwelling older adults for two months; the comparison group provided their routine services at senior activity centers. Data were collected at baseline, one month, and three months into the study.

ELIGIBILITY:
Inclusion Criteria:

* older adults age ≥ 65
* able to read and write in Chinese
* being a volunteer at the senior activity center for at least 1 month

Exclusion Criteria:

* illiterate

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 162 (Actual)
Dates: Start 2023-06-16 (Actual); Primary Completion 2023-12-08 (Actual); Study Completion 2023-12-08 (Actual)

PRIMARY OUTCOMES:
knowledge and skills of volunteer work | 3 months
  measured by the Older Volunteer Competency Scale. It has 30 items with 3 sub-scales. Each item is measured by a 10-point Likert scale. The item scores represent the perceived improvement needed by the respondents with higher scores indicating more needed improvements.

SECONDARY OUTCOMES:
motivation for volunteering | 3 months
  measured by the Volunteer Functions Inventory. It contains 30 items in 6 sub-scales to assess volunteers' motivational functions. Each item is rated on a 7-point Likert scale. A higher score indicates a greater importance of that motive.
self-efficacy | 3 months
  measured by the Volunteers' Self-efficacy Questionnaire. It contains 25 items measuring four dimensions. Each item is rated on a 5-point Likert scale. A higher score indicates better self-efficacy.
satisfaction with volunteer work | 3 months
  measured by the Working Satisfaction Scale. It is comprised of 13 items assessing 3 dimensions. Each item is rated on a 5-point Likert scale. A higher score indicates higher satisfaction with volunteer work.

CONTACTS AND LOCATIONS:
Overall Officials: Kuei-Min Chen, PhD, Principal Investigator — Kaohsiung Medical University, Taiwan
Locations (1):
- Kaohsiung Medical University, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No